CLINICAL TRIAL: NCT06030960
Title: The Effects of Virtual Reality Stabilization Training on Postural Stability and Proprioception in Patients With Low Back Pain
Brief Title: Effects of Virtual Reality Stabilization Training in Patients With Low Back Pain
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Abrar AlSadiq, Rehabilitation Sciences PhD Student, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2023-03-097
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: LBP; Psychological effects; Intervention; Virtual Reality; postural stability; balance; pain; COP
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients with Chronic Low Back Pain (CLBP) who will receive Virtual Reality (VR) stabilization exercises, regular stabilization exercises and patient instructions and education
  Interventions: Device: Virtual Reality (VR); Other: Regular Exercises; Other: patient instructions and education
- Group 2 (Active Comparator): Patients with Chronic Low Back Pain (CLBP) who will receive regular stabilization exercises and patient instructions and education
  Interventions: Other: Regular Exercises; Other: patient instructions and education

INTERVENTIONS:
Device: Virtual Reality (VR) — Virtual Reality (VR) Stabilization Exercises
  Other Names: Exergames
  Arms: Group 1
Other: Regular Exercises — Regular Stabilization Exercises
Other: patient instructions and education — a unified form of patient instructions and education in regards of LBP

SUMMARY:
To our knowledge, no studies have better investigated the effect of Core Stabilization Exercises using VR on ankle and trunk proprioception in patients with CLBP and in turn on postural stability.

DETAILED DESCRIPTION:
Background: Low Back Pain (LBP), one of the most critical disability causatives, has been associated with neuromuscular and biomechanical manifestations related to the deficiency of postural control and stability. Virtual reality (VR) core stabilization exercises (CSE) has proven previously to be effective in improving postural control among conditions with different proprioceptive damage mechanisms other than those affected with LBP. The Aim of this study is to explore the differing effects of this treatment regimen on postural stability in relation to lumbar and ankle proprioception in a population of participants with LBP. Design and Methods: a randomized clinical trial encompassing 44 participants of both genders. Participants with Chronic Low Back Pain (CLBP) will be randomized to one of two treatment groups: an Experimental group receiving VR stabilization exercises and a Control group receiving CSE only without VR simulations inaddition to patient instructions and education of both groups. Parameters of postural stability, ankle and trunk proprioception, pain intensity, balance interference with activity and psychological aspects of pain interference with activity will be measured by a force plate, iPhone applications, visual analog scale (VAS), the Activities-specific Balance Confidence (ABC) scale, Pain Catastrophizing Scale (PCS) and the Pain Self-Efficacy Questionnaire (PSEQ-Ar) respectively. Outcome measures will be collected at baseline, immediately after 1st treatment and after the last treatment session. Treatment regimens will consist of 12 sessions in 3 weeks using virtual reality glasses. Statistical Analysis: A linear mixed model will be used to analyze within- and between-group differences at the baseline, 6th session and twelfth sessions (repeated measures will be set as GROUP with two levels and TIME with three levels). Bonferroni post-hoc procedures will be used for multiple comparisons of the differences over time. Intention-to-treat analysis shall be utilized. Statistical significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients in Group 1 and Group 2 will be included if they:

1. Are adults between 25 and 59 years of age.
2. Have LBP for longer than 3 months.
3. Are not currently undergoing medication or conservative treatment.

Exclusion Criteria:

Patients in these two groups will be excluded if they have:

1. Nerve root manifestations (such as referred symptoms of radiating pain below the knee or paresthesia during the straight leg raise test),
2. Systematic or visceral disease,
3. Ankylosing spondylitis, Spondylolysis and Spondylolisthesis,
4. Vestibular dysfunctions,
5. Body mass index (BMI) ≥ 30 kg/m2,
6. Lower extremity injury within the past month,
7. Concussion,
8. Psychiatric, cardiovascular or musculoskeletal disorders,
9. Vision problems,
10. Vertebral fracture,
11. Spinal Stenosis,
12. Previous spinal surgery,
13. Present pregnancy,
14. Scoliosis,
15. Inability to understand instructions, read or write (Li et al., 2021).

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Postural stability | 12 weeks
  Centre of Pressure (CoP) movements will be tracked by a multi-sensory platform + Body Weight Balance (static):
Proprioception | 12 weeks
  Ankle and Trunk Joint Position Sense (JPS)

SECONDARY OUTCOMES:
Pain Intensity | 12 weeks
  Visual Analog Scale (VAS)
Pain Self-Efficacy Questionnaire (PSEQ-Ar) | 12 weeks
  to examine one's beliefs, level of Pain intensity and actual achievements contributions to performance
Activities-specific Balance Confidence (ABC) | 12 weeks
  Active clinical assessment measures of balance and function
Pain Catastrophizing Scale | 12 weeks
  Overstressed undesirable perceptions of pain and the ambiance surrounding its involvement

CONTACTS AND LOCATIONS:
Overall Officials: Ali AlShami, PhD, Study Chair — alshami@iau.edu.sa
Locations (1):
- Dammam Medical Complex, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No